CLINICAL TRIAL: NCT02919436
Title: Decreasing Rates of Intraurethral Catheterization Postoperatively in Spine Surgery
Acronym: DRIPS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Anand Rughani, MD (Other)
Collaborators: MaineHealth (Other)
Responsible Party: Sponsor-Investigator, Anand Rughani, MD, Neurosurgeon, MaineHealth
Organization: MaineHealth (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB #4742
Record Dates: First submitted 2016-09-28; First posted 2016-09-29 (Estimated); Results first posted 2022-02-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-01

CONDITIONS: Post-operative Urinary Retention
MeSH Terms: interventions — Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tamsulosin (Experimental): Subjects in this arm will receive tamsulosin 0.4 mg/day for five days prior to surgery and two days after surgery.
  Interventions: Drug: Tamsulosin
- Placebo (Placebo Comparator): Subjects in this arm will receive a placebo capsule identical in appearance to the tamsulosin capsule, for five days prior to surgery and two days after surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tamsulosin — Active drug
  Other Names: Flomax; Flomaxtra; Contiflo XL; Urimax
  Arms: Tamsulosin
Drug: Placebo — Lactose-filled capsules identical to active drug
  Arms: Placebo

SUMMARY:
Randomization (1:1) of male patients, over age 50, undergoing elective spine surgery to tamsulosin versus a placebo.

DETAILED DESCRIPTION:
Postoperative urinary retention (POUR) is a common complication following certain surgical operations. While much is known about the innervation and neural regulation of bladder emptying and storage, the cause of urinary retention after surgery is not fully understood. Early research has indicated that a small dose of tamsulosin (Flomax®), a commonly used medication approved to treat urinary symptoms in men with benign prostatic hypertrophy, may reduce the incidence of POUR. Urinary retention is a prevalent issue in patients undergoing spinal surgery, leading to patient discomfort and prolonged length of stay. We hypothesize that the use of perioperative tamsulosin in patients undergoing spinal surgery will decrease the incidence of POUR.

The study is a prospective, double-blind, randomized, placebo-controlled trial. Subjects will be randomized 1:1 to receive either oral tamsulosin 0.4 mg or placebo, taken once each evening, beginning 5 days prior to surgery and continuing through the first postoperative day. The primary endpoint is met when the patient is able to spontaneously empty their bladder post-operatively, or needs to be catheterized with either a straight or indwelling urinary catheter for post-operative urinary retention, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria

* Male patient age 50 - 85 years
* Undergoing elective spine surgery at least 5 days after enrollment
* Preop visit done at office practice

Exclusion Criteria:

* Currently on tamsulosin or other alpha-adrenergic blocking drug
* Allergy to tamsulosin
* Allergy to lactose
* Serious or life-threatening allergy to sulfa drugs
* Emergent procedure
* History of spinal trauma, spinal infection or spinal cord tumor
* Pre-existing indwelling urinary catheter
* History of orthostatic hypotension or current orthostatic hypotension
* History of prostate, urethral or bladder surgery
* Renal failure
* Non-English speaking
* Unable to provide informed consent

Ages: 50 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 610 (Actual)
Dates: Start 2016-03; Primary Completion 2020-01 (Actual); Study Completion 2020-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anand Rughani, MD, Principal Investigator — MaineHealth
Locations (1):
- Maine Medical Center, Portland, Maine, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible subjects were enrolled at a neurosurgery outpatient clinic from 2016 to 2019, and included males age 50 to 85 undergoing elective spine surgery at least 5 days after study enrollment.
Pre-assignment Details: Patients not enrolled included those who did not meet entry criteria (n=150), those who declined to participate (n=140) and those who were not enrolled for other reasons (n=151).
Period: Overall Study
Arm/Group | Tamsulosin | Placebo
Started | 305 | 305
Completed | 245 | 252
Not Completed | 60 | 53
Not completed — Did not undergo surgery | 16 | 20
Not completed — Enrolled before trial registration | 44 | 33

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tamsulosin | Placebo | Total
Number analyzed (Participants) | 245 | 252 | 497
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (7.7) | 63.7 (8.7) | 63.5 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 245 | 252 | 497
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
History of hypertension [Count of Participants; unit: Participants] | 165 | 163 | 328
History of insulin-dependent diabetes mellitus [Count of Participants; unit: Participants] | 21 | 19 | 40
History of non-insulin dependent diabetes mellitus [Count of Participants; unit: Participants] | 59 | 49 | 108
History of benign prostatic hyperplasia [Count of Participants; unit: Participants] | 15 | 23 | 38
Current opioid use [Count of Participants; unit: Participants] | 55 | 52 | 107
Current smoker [Count of Participants; unit: Participants] | 48 | 36 | 84
Body mass index > 30 [Count of Participants; unit: Participants] | 130 | 136 | 266
BMI mean [Mean (Standard Deviation); unit: kg/m^2] | 30.9 (5.7) | 31.1 (5.6) | 31.1 (5.6)
Office post-void residual < 50 cc [Count of Participants; unit: Participants] — Measurement by ultrasound of the amount of urine remaining in bladder after urinating
  Participants | 141 | 150 | 291
Modified International Prostate Symptom Score mean [Mean (Standard Deviation); unit: Scores on a scale] — Scale measures clinical symptoms of prostate enlargement, with range of 0 (no symptoms) to 25 (severe symptoms).
  Scores on a scale | 5.1 (4.6) | 4.9 (4.2) | 5.0 (4.4)
Lumbar spine surgery [Count of Participants; unit: Participants] | 175 | 199 | 374
Arthrodesis performed [Count of Participants; unit: Participants] | 66 | 62 | 128

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Undergo Postoperative Catheterization for Urinary Retention
Description: Postoperative urinary retention was defined as the need for any postoperative urinary catheterization for acute retention. Per hospital protocol, failure to void 6 hours after surgery or development of bladder discomfort required bladder scan. If bladder volume exceeded 300 cc, catheterization was performed.
Time Frame: Within 2 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Tamsulosin | Placebo
Number analyzed (Participants) | 245 | 252
Participants | 23 | 25
Statistical Analysis 1: Comparison: Tamsulosin vs Placebo; Test type: Superiority — We found observed rate of postoperative urinary retention in male spine surgery patients to historically be 17%. We hypothesize that the use of tamsulosin can reduce this rate by 50%. A two group continuity corrected chi-square test with a .05 two-sided significance level will have 80% power to detect the difference between a control group proportion of .17 and a treatment group proportion of .085 (odds ratio of .454) when the sample size in each group is 264 and a total sample size of 528; p = .96, Chi-squared, Corrected

2. Secondary Outcome: Length of Stay
Description: Length of hospital stay
Time Frame: 0-7 days after surgery
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tamsulosin | Placebo
Number analyzed (Participants) | 245 | 252
days | 0.9 (1.2) | 0.7 (0.9)

3. Secondary Outcome: Number of Participants With or Without Postoperative Urinary Retention Based on Preoperative Post-void Residual
Description: Was post-void residual greater than 50 cc when measured at the preoperative office visit associated with postoperative urinary retention?
Time Frame: Within 2 days after surgery
Population: Overall number of participants analyzed in this section (447) is different than total number analyzed overall (497), because PVR was a missing value on 50 patients. This was due to bladder scanner used to measure PVR being inoperable several times over the course of the study.
Measure: Count of Participants; unit: Participants
Groups:
- Preoperative Post-void Residual < 50 cc: Subjects in this group had a post-void residual greater than 50 cc in the preoperative office visit
- Preoperative Post-void Residual >/= 50 cc: Subjects in this group had a post-void residual greater than or equal to 50 cc in the preoperative office visit
Arm/Group | Preoperative Post-void Residual < 50 cc | Preoperative Post-void Residual >/= 50 cc
Number analyzed (Participants) | 291 | 156
Participants
  Postoperative urinary retention | 18 | 22
  No postoperative urinary retention | 273 | 134

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 2 weeks following each subject's discharge from the hospital.
Arm/Group | Tamsulosin | Placebo
All-Cause Mortality (participants affected / at risk) | 1/245 | 0/252
Serious Adverse Events (participants affected / at risk) | 5/245 | 4/252
Other Adverse Events (participants affected / at risk) | 25/245 | 15/252
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tamsulosin (N=245) | Placebo (N=252)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 2 (2) | 1 (1)
Postop neurosurgical complication (Surgical and medical procedures) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Other (General disorders) | 0 (0) | 2 (2) — C. difficile encephalopathy (1) and Urosepsis (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tamsulosin (N=245) | Placebo (N=252)
Urinary issues (Renal and urinary disorders) | 7 (7) | 8 (8) — Includes urinary frequency, dribbling, difficulty voiding
Nausea / emesis (Gastrointestinal disorders) | 5 (5) | 1 (1)
Headache (General disorders) | 3 (3) | 0 (0)
Cardiac (Cardiac disorders) | 1 (1) | 1 (1)
Other (General disorders) | 9 (9) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-03): https://cdn.clinicaltrials.gov/large-docs/36/NCT02919436/Prot_SAP_000.pdf